CLINICAL TRIAL: NCT05151393
Title: Correlation Between Serum Vitamin D3 Level and Incidence of Uterine Leiomyoma in Egyptian Women
Brief Title: Correlation Between Serum Vitamin D3 and Incidence of Uterine Leiomyoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed Samy, Obs/Gyn resident, Ain Shams University
Other Study IDs: VitaminD and Uterine leiomyoma
Record Dates: First submitted 2021-08-24; First posted 2021-12-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: Vitamin D Deficiency; Leiomyoma
MeSH Terms: conditions — Vitamin D Deficiency; Leiomyoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Cases with uterine leiomyoma
  Interventions: Diagnostic Test: Measuring vitamin D3 level
- Controls: Cases free of uterine leiomyoma
  Interventions: Diagnostic Test: Measuring vitamin D3 level

INTERVENTIONS:
Diagnostic Test: Measuring vitamin D3 level — Measuring vitamin D3 in both groups

SUMMARY:
The aim of the current study is to evaluate the association between low serum vitamin D level and incidence of uterine leiomyoma in Egyptian women as the research hypothesis that low serum vitamin D is considered a risk factor for uterine leiomyoma

ELIGIBILITY:
Inclusion Criteria:

1. Age ranging from 20 to 45 years.
2. Postmenstrual patients to exclude current pregnancy.
3. Parity up to para 3 by either normal vaginal delivery or cesarean section.
4. Body mass index (BMI) ranging from 18 to 30 kg/m2.
5. One or more uterine fibroid with a diameter ranging from 3-10 cm.
6. Fibroids either subserous, intramural or submucous uterine fibroids

Exclusion Criteria:

1. Women aged less than 20 years have a very low incidence of fibroids or more than 45 years as there is an increased incidence of vitamin D deficiency after this age.
2. Patients known to be currently pregnant due to change in fibroids volume during pregnancy in addition to vitamin D levels may be lower than baseline for nonpregnant ones.
3. Grand multipara >3 times frequently associated with vitamin D deficiency.
4. Cardiac( e.g rheumatic heart diseases), pulmonary( e.g asthma, bronchiectasis ), or hematological disease (including anemia; hemoglobin level below 10gm/dl , thalassemia, sickle cell anemia, and spherocytosis) because of high association between chronic illnesses and multivitamin deficiency.
5. Patients who receive pre-operative hormonal therapy (such as GnRH analogue) which may increase vitamin D levels and interfere with the study objectives.
6. Patients who will present with a suspected malignant gynecological disease which is usually associated with multiple vitamin deficiencies including vitamin D.
7. Patients who will be diagnosed as having cervical or supracervical fibroids and pedunculated fibroids (study will be limited on corporeal fibroid).
8. Small fibroid less than 3cm diameter may not be enough size to cause changes in lab results or large ones more than 10 cm diameter.
9. Previous myomectomy or hysterectomy.
10. Using vitamin supplements or hormonal therapy during or within 6 months of enrolment which may interfere with the accurate results of the study.
11. Current lactating or lactating within 6 months prior to enrollment as breastfeeding women have a significantly higher prevalence of vitamin D deficiency.
12. Current smokers or history of smoking as it decreases the production of the active form of vitamin D.
13. Steroids intake as it increases the 24-hydroxylase level causing vitamin D deficiency.
14. Cases diagnosed with any form of malignancy that may be associated with vitamin D deficiency.
15. Current treatment with heparin as it interferes with vitamin D activation.
16. Patients currently on depo-medroxyprogesterone-acetate (DMPA) contraceptives as it proved benefits in shrinking fibroid size.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Study Population: (N=80) Women with symptomatic uterine fibroids attending the gynecology outpatient clinic and age matched controls free from uterine leiomyoma.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-01-28 (Estimated); Study Completion 2022-02-15 (Estimated)

PRIMARY OUTCOMES:
Low levels serum vitamin D as a risk factor for development of uterine leiomyoma. | 6 months
  Low levels serum vitamin D as a risk factor for development of uterine leiomyoma.

SECONDARY OUTCOMES:
Correlation of low serum vitamin D with size, site and number of fibroids | 6 months
  Correlation of low serum vitamin D with size, site and number of fibroids
Correlation of low serum vitamin D with severity of symptoms related to uterine leiomyoma | 6 months
  Correlation of low serum vitamin D with severity of symptoms related to uterine leiomyoma
Role of vitamin D deficiency in development of uterine leiomyoma in high risk groups (black race, obese patients). | 6 months
  Role of vitamin D deficiency in development of uterine leiomyoma in high risk groups (black race, obese patients).

CONTACTS AND LOCATIONS:
Overall Officials: Rania Gamal, MD, Study Director — Ain Shams University; Mortada Elsayed, MD, Study Director — Ain Shams University; Aliaa Maaty, MD, Study Director — Ain Shams University; Magdy Hassan, MD, Study Chair — AinShansU

REFERENCES:
- [Background] Corachan A, Ferrero H, Escrig J, Monleon J, Faus A, Cervello I, Pellicer A. Long-term vitamin D treatment decreases human uterine leiomyoma size in a xenograft animal model. Fertil Steril. 2020 Jan;113(1):205-216.e4. doi: 10.1016/j.fertnstert.2019.09.018. Epub 2019 Nov 15. PMID 31739978
- [Background] Bouillon R, Carmeliet G. Vitamin D insufficiency: Definition, diagnosis and management. Best Pract Res Clin Endocrinol Metab. 2018 Oct;32(5):669-684. doi: 10.1016/j.beem.2018.09.014. Epub 2018 Oct 3. PMID 30449548
- [Background] Ciavattini A, Clemente N, Delli Carpini G, Di Giuseppe J, Giannubilo SR, Tranquilli AL. Number and size of uterine fibroids and obstetric outcomes. J Matern Fetal Neonatal Med. 2015 Mar;28(4):484-8. doi: 10.3109/14767058.2014.921675. Epub 2014 Jun 5. PMID 24803127
- [Background] Ciebiera M, Ali M, Zgliczynska M, Skrzypczak M, Al-Hendy A. Vitamins and Uterine Fibroids: Current Data on Pathophysiology and Possible Clinical Relevance. Int J Mol Sci. 2020 Aug 1;21(15):5528. doi: 10.3390/ijms21155528. PMID 32752274
- [Background] Drayer SM, Catherino WH. Prevalence, morbidity, and current medical management of uterine leiomyomas. Int J Gynaecol Obstet. 2015 Nov;131(2):117-22. doi: 10.1016/j.ijgo.2015.04.051. Epub 2015 Aug 5. PMID 26275638
- [Background] Mas A, Tarazona M, Dasi Carrasco J, Estaca G, Cristobal I, Monleon J. Updated approaches for management of uterine fibroids. Int J Womens Health. 2017 Sep 5;9:607-617. doi: 10.2147/IJWH.S138982. eCollection 2017. PMID 28919823
- [Background] Mettler L, Schollmeyer T, Tinelli A, Malvasi A, Alkatout I. Complications of Uterine Fibroids and Their Management, Surgical Management of Fibroids, Laparoscopy and Hysteroscopy versus Hysterectomy, Haemorrhage, Adhesions, and Complications. Obstet Gynecol Int. 2012;2012:791248. doi: 10.1155/2012/791248. Epub 2012 Apr 9. PMID 22619681
- [Background] Matsui MS. Vitamin D Update. Curr Dermatol Rep. 2020;9(4):323-330. doi: 10.1007/s13671-020-00315-0. Epub 2020 Oct 14. PMID 33078087
- [Background] Sheng B, Song Y, Liu Y, Jiang C, Zhu X. Association between vitamin D and uterine fibroids: a study protocol of an open-label, randomised controlled trial. BMJ Open. 2020 Nov 6;10(11):e038709. doi: 10.1136/bmjopen-2020-038709. PMID 33158822
- [Background] Singh V, Barik A, Imam N. Vitamin D3 Level in Women with Uterine Fibroid: An Observational Study in Eastern Indian Population. J Obstet Gynaecol India. 2019 Apr;69(2):161-165. doi: 10.1007/s13224-018-1195-4. Epub 2018 Dec 6. PMID 30956471
- [Background] Sirajudeen S, Shah I, Al Menhali A. A Narrative Role of Vitamin D and Its Receptor: With Current Evidence on the Gastric Tissues. Int J Mol Sci. 2019 Aug 5;20(15):3832. doi: 10.3390/ijms20153832. PMID 31387330
- [Background] Srivastava P, Gupta HP, Singhi S, Khanduri S, Rathore B. Evaluation of 25-hydroxy vitamin D3 levels in patients with a fibroid uterus. J Obstet Gynaecol. 2020 Jul;40(5):710-714. doi: 10.1080/01443615.2019.1654986. Epub 2019 Oct 22. PMID 31635506
- [Background] Stewart EA, Cookson CL, Gandolfo RA, Schulze-Rath R. Epidemiology of uterine fibroids: a systematic review. BJOG. 2017 Sep;124(10):1501-1512. doi: 10.1111/1471-0528.14640. Epub 2017 May 13. PMID 28296146
- [Background] Szkodziak P, Pyra K, Szkodziak F, Krzyzanowski J, Czuczwar P, Wozniak S, Jargiello T, Paszkowski T. The Lublin Protocol of the Uterine Arteries Embolization in the Treatment of Symptomatic Uterine Fibroids. J Vis Exp. 2020 Sep 15;(163). doi: 10.3791/61530. PMID 33016950